CLINICAL TRIAL: NCT01198210
Title: Comparison of Peritonsillar Infiltration of Ketamine and Dexamethasone for Postoperative Pain Relief in Children Following Adenotonsillectomy
Brief Title: The Effect of Peritonsillar Infiltration of Ketamine and Dexamethasone for Postoperative Pain Relief in Children Following Adenotonsillectomy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, marzieh beigom khezri, Assistant professor, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ACTRN12610000658011
Record Dates: First submitted 2010-09-01; First posted 2010-09-10 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Tonsillectomy
Keywords: pain; tonsillectomy; peritonsillar infiltration; postoperative pain
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Sodium Chloride; Ketamine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- saline (Placebo Comparator): One hundred sixtyAmerican Society of Anesthesiologists (ASA) I-II children 3-12 were randomized four groups of 40 each. Group P received a local peritonsillar infiltration of 2 ml saline, group D dexamethsone (0.2 mg/kg)) , group K ketamine (0.5 mg/kg) and group KD combination of ketamine0.5mg/kg-dexamethasone 0.2mg/kg. All medications were 2 ml in volume which was applied 1 ml per tonsil 3 min prior to tonsillectomy( all four groups).
  Interventions: Drug: saline
- ketamine (Active Comparator): One hundred sixtyAmerican Society of Anesthesiologists (ASA) I-II children 3-12 were randomized four groups of 40 each. Group P received a local peritonsillar infiltration of 2 ml saline, group D dexamethsone (0.2 mg/kg)) , group K ketamine (0.5 mg/kg) and group KD combination of ketamine0.5mg/kg-dexamethasone 0.2mg/kg. All medications were 2 ml in volume which was applied 1 ml per tonsil 3 min prior to tonsillectomy( all four groups).
  Interventions: Drug: Ketamine
- dexamethasone (Active Comparator): One hundred sixtyAmerican Society of Anesthesiologists (ASA) I-II children 3-12 were randomized four groups of 40 each. Group P received a local peritonsillar infiltration of 2 ml saline, group D dexamethsone (0.2 mg/kg)) , group K ketamine (0.5 mg/kg) and group KD combination of ketamine0.5mg/kg-dexamethasone 0.2mg/kg. All medications were 2 ml in volume which was applied 1 ml per tonsil 3 min prior to tonsillectomy( all four groups).
  Interventions: Drug: Dexamethasone
- dexamethasone-ketamine (Active Comparator): One hundred sixtyAmerican Society of Anesthesiologists (ASA) I-II children 3-12 were randomized four groups of 40 each. Group P received a local peritonsillar infiltration of 2 ml saline, group D dexamethsone (0.2 mg/kg)) , group K ketamine (0.5 mg/kg) and group KD combination of ketamine0.5mg/kg-dexamethasone 0.2mg/kg. All medications were 2 ml in volume which was applied 1 ml per tonsil 3 min prior to tonsillectomy( all four groups).
  Interventions: Drug: ketamine-dexamethasone

INTERVENTIONS:
Drug: saline — local peritonsillar infiltration of 2 ml saline,
  Arms: saline
Drug: Ketamine — local peritonsillar infiltration of ketamine (0.5 mg/kg)
  Arms: ketamine
Drug: Dexamethasone — local peritonsillar infiltration dexamethasone (0.2 mg/kg))
  Arms: dexamethasone
Drug: ketamine-dexamethasone — local peritonsillar infiltration combination of ketamine0.5mg/kg-dexamethason 0.2mg/kg
  Arms: dexamethasone-ketamine

SUMMARY:
The immediate postoperative period after tonsillectomy, , is often difficult. These children frequently have severe pain but postoperative airway edema along with increased sensitivity to the respiratory-depressant effects of opioids may result in obstructive symptoms and hypoxemia. Opioid consumption may be reduced by non-steroidal anti-inflammatory drugs, but these drugs may be associated with increased bleeding after this operation.

Methods: One hundred sixty ASA I-II children 3-12 were randomized four groups of 40 each. Group P received a local peritonsillar infiltration of 2 ml saline, group D dexamethsone (0.2 mg/kg)) , group K ketamine (0.5 mg/kg) and group KD combination of ketamine0.5mg/kg dexamethasone 0.2mg/kg. All medications were 2 ml in volume which was applied 1 ml per tonsil 3 min prior to tonsillectomy. Study drugs were marked only with a coded number label. A computer-generated table of numbers guided randomization. Modified Hannallah pain scale [observational pain scores (OPS)], nausea, vomiting, bleeding, rescue analgesia, sedation and Aldrete scores were recorded at first, 15th, 30th and 60th min postoperatively. Patients were interviewed on the day after surgery to assess the postoperative pain, nightmares, hallucinations, vomiting and bleeding. All the children were premedicated with midazolam hydrochloride 0.3 mg/kg) and fentanyl 1micro g/kg intavenously. Anesthesia was induced with thiopental 5mg/kg and atracurium0.3mg/kg. Anesthesia was maintained with isoflurane 1.5% and nitrous oxide 30% in oxygen. The two surgeon used the same dissection and snare technique for all cases and hemostasis done with bipolar cutter. At the end of the surgery neuromuscular blockade was reversed by neostigmine 0.03 mg/kg) and atropine 0.01 mg/kg intravenously), anesthesia was discontinued and the tracheal tube removed in the operating room when patients were deep. After extubation the patients were taken to the postanesthesia care unit (PACU) where an nurse who were unaware of the study drug observed the patients. The pain scoring observer nurse in PACU was consistent. Time to awaken (from the end of anesthesia until the patients opened their eyes on command) and time to the first administration of postoperative analgesia were recorded. Pethidine in a titrated dose (total 1 mg/kg) was administered intravenously for rapid pain relief to patients with a OPS score > 4 or who were crying during two consecutive five minute observation periods until the child was comfortable. Postoperative pain during the first 24 h was assessed using a four-point scale: 0 no pain, 1 mild pain, 2 moderate pain, 3 severe pain by questioning their parents. In the ward the standardized postoperative analgesic technique was with acetaminophen supp (40 mg/kg followed by three doses of 20 mg/kg at 6-hour intervals to be given as needed for pain. Pethidine in a titrated dose (total 1 mg/kg) was administered intravenously for rapid pain relief to patients who had pain scale >3.Any supplementary analgesia , nausea and vomiting, bleeding, sleep disturbance and nightmares that the child might have had as surgery were assessed during a telephone follow up 24 h later.

ELIGIBILITY:
Inclusion Criteria:

* children age 3-12 years ASAI,II

Exclusion Criteria:

* contraindication for usage of Ketamine, dexamethasone
* upper respiratory tract infection
* increase intracranial pressure( ICP)
* history of allergy ,seizure,psychiatric illness, , bleeding disorders
* chronic usage of analgesic ,antiemetic ,stroied drugs two weeks before surgery,
* history of peritonsillar abscess, , tonsillitis within two weeks, -

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
pain will be assessed by [observational pain scores (OPS)] | 5 minutes After extubation when the patients were taken to the postanesthesia care unit (PACU)
pain will be assessed by [observational pain scores (OPS)] | 15th min postoperatively (15 minutes After extubation when the patients were taken to the postanesthesia care unit (PACU))
pain will be assessed by [observational pain scores (OPS)] | 30th min postoperatively (30 minutes After extubation when the patients were taken to the postanesthesia care unit (PACU))
pain will be assessed by [observational pain scores (OPS)] | 60thmin postoperatively (60 minutes After extubation when the patients were taken to the postanesthesia care unit (PACU))
time to first demand of analgesia | during 60min postoperatively (during 60 minutes After extubation when the patients were taken to the postanesthesia care unit (PACU))
postoperative analgesic consumption | during 24 h postoperative (in the ward)

SECONDARY OUTCOMES:
nausea, vomiting will be assessed by questioning their parents. | during 60th min after extubation at postanesthesia care unit
bleeding will be assessed by questioning their parents | during 24 h postoperative (in the ward)
family satisfaction will be assessed by questioning their parents. | during 24 h postoperative (in the ward).
nausea, vomiting will be assessed by questioning their parents. | during 24 h postoperative (in the ward)

CONTACTS AND LOCATIONS:
Locations (1):
- Qazvin university of medical science, Qazvin, Qazvin Province, Iran